CLINICAL TRIAL: NCT05825170
Title: A Prospective Clinical Investigation Evaluating the Safety and Effectiveness of FASY L Hyaluronic Acid Gel for the Treatment of Lip Deformity
Brief Title: Evaluation of a HA Dermal Filler in the Treatment of Lip Deformity
Acronym: FENTHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Symatese (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN2202
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Lip, Cleft; Lip Scar
Keywords: Hyaluronic acid; Dermal fillers; lips
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FASY L (Experimental): Subjects will be consecutively included to receive FASY L in lips at level of their scar
  Interventions: Device: FASY L

INTERVENTIONS:
Device: FASY L — Subjects will receive FASY L in lips at level of their scar.

SUMMARY:
Early postnatal repair of cleft lip and palate aims at the development of the child through reconstruction of the face soon after birth. Cleft lip is the result of a defect in the fusion of the buds of the face by default of cell apoptosis of the embryonic neural crest constituting the skin and the labial mucosa. Lip surgery or cheiloplasty primary of unilateral and bilateral cleft lip and palate is carried out from the age of 6 weeks. At the end of the surgical treatment, we often observe small unsightly residual volumetric asymmetries. The choice is then either to surgically reduce a muscular part too voluminous by reducing locally the volume of the lip, or to increase the volume of the thinnest portion this second solution is made possible either by injecting fat or by injection of hyaluronic acid. By adulthood, patients with cleft lip have often undergone 10 or more defect-related surgeries and many desire less invasive options to improve any residual cosmetic imperfections. The first use of a temporary alloplastic injectable soft tissue filler, hyaluronic acid (HA), for upper lip augmentation in a patient with asymmetry after surgical cleft lip repair was reported in 2008. There are few publications on the use hyaluronic acid in complement to the surgical treatment of cleft lip and palate, but all reported promising results.

DETAILED DESCRIPTION:
The study is a pilot, prospective, multicenter, proof-of-concept clinical trial that aims to evaluate the safety and efficacy of FASY L for the treatment of lip deformity.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female.
* Age: 18 years and older.
* Women of childbearing age must have a negative urine pregnancy test before each injection.
* Patient seeking an enhancement of the lip deformity with FASY L after having undergone cleft lip and palate surgical treatment.
* Patient, having given freely and expressly his/her informed consent.
* Patient who is able to comply with the study requirements, as defined in the present CIP, at the Investigator's appreciation.
* Patient being affiliated to a health social security system.

Exclusion Criteria:

* Pregnant and breastfeeding women
* Subject who is deprived of their freedom by administrative or legal decision.
* Subject living in a social or sanitary establishment.
* Major subject who is under guardianship or who is not able to express his consent.
* Subject being in an exclusion period for a previous study or with a current or recent (<3 months) participation in another investigational study involving a drug or combined device with drug.
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results: diabetes, autoimmune pathology, cardiac pathologies, hepatic deficiency, epilepsy, porphyria.
* Subject who has a known history of severe multiple allergies, angioedema or anaphylactic shock.
* Subject with a known allergy or hypersensitivity to Hyaluronic Acid or local anesthesia (Lidocaine or anesthetics of the amide type or any of the excipients).
* Subject with an acute inflammatory process or active skin disease, or related conditions, such as infection, psoriasis, rosacea, acne, blotches or other pathology near or on the injection sites with the potential to interfere with the study results or increase the risk of Adverse Events at the Investigator appreciation.
* Subject with a past history of severe streptococcal disease or an active streptococcus infection.
* Subject predisposed to keloid or hypertrophic scarring.
* Subject with a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder.
* Subject with a history of precancerous lesions/skin malignancies on the injection sites.
* Subject with history of hyper- or hypo-pigmentation on the face.
* Subject with a known bleeding disorder or receiving medication that will likely increase the risk of bleeding during treatment, at the Investigator appreciation.
* Subject having received high dose of Lidocaine (more than 200mg) and/or high dose of anesthetics structurally related to amide-type within the past week.
* Subject having received chemotherapy agents, immunosuppressive medications or systemic corticosteroids within the past 3 months.
* Patient having taken high-dose aspirin, anti-inflammatories, antiplatelet, thrombolytic during the week before the injection session.
* Subject having received within the past 12 months any injections including non-permanent fillers (e.g., Hyaluronic Acid, CaHA), mesotherapy or neurotoxin near or on the lips or plan to undergo such treatment during the study.
* Subject with prior permanent implant or treatment with non-HA or non-collagen filler near or on the lip or plan to implement these products at any time during the study.
* Subject having received within the past 6 months mesotherapy, resurfacing laser, photo modulation, intense pulsed light, radio frequency, photo-rejuvenation, dermabrasion, chemical peel, or other ablative or none ablative procedures near or on the lips.
* Subject with subcutaneous retaining structure on the face (meshing, threads, gold strand etc.) near or on the injection sites (lips) with the potential to interfere with the study results or increase the risk of Adverse Events at the Investigator appreciation.
* Patient having received fat grafting within the past 6 months near or on the injection sites
* Other condition preventing the subject to participate the study in the Investigator's opinion: subject deemed unreliable or incapable of understanding and complying with the study assessment or unrealistic expectations of treatment results.
* Subject who planned an intensive exposure to sunlight or UV-rays in the 2 weeks following injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with at least one Adverse Device Event (ADE) at the visit at 30 days after the initial injection | 30 days visit after the first injection
  Recording of the occurrence of Adverse Event related to the use of the investigational medical device. Assessed by investigators.

SECONDARY OUTCOMES:
Injection Site Reactions present immediatly after injections | Day 0 and potentially at each visits (Day 30, Month 3, Month 6, Month 9 and Month 12 after the first injection)
  Recording of the presence and severity (mild, moderate or severe) of local injection site reactions after each injection.
Evaluation of the scar by the investigators | Before the first injection (baseline) and Day 30, Month 3, Month 6, Month 9 and Month 12 after the first injection
  Assessement of the scar using the Patient and Observer Scar Assessment Scale (POSAS).
  The POSAS of the observer includes six parameters (vascularity, pigmentation, thickness, relief, elasticity and surface). In addition, a general opinion is scored. Each parameter is rated by the investigator on a scale from 1 ("normal skin") to 10 ("worst scar imaginable"). The sum of the seven parameters constitutes the total score of the scale of the observer ranging from 7 (normal skin) to 70 (worst scar imaginable).
Evaluation of the scar by the patients | Before the first injection (baseline) and Day 30, Month 3, Month 6, Month 9 and Month 12 after the first injection
  Assessement of the scar using the Patient and Observer Scar Assessment Scale (POSAS).
  The POSAS ot the patient includes six questions about pain, itching, color, roughness, thickness and irregularities of the scar. In addition, a general opinion is scored. Each parameter is rated by the patient on a scale from 1 ("no, not at all") to 10 ("yes, extremely"). The sum of the seven parameters constitutes the total score of the scale of the patients ranging from 7 (normal skin) to 70 (worst scar imaginable)..
Incidence of Treatment-Emergent Adverse Events | Day 30, Month 3, Month 6, Month 9 and Month 12 after the first injection.
  Collection of Adverse Event assessed and recorded by investigators.
Patient Global aesthetic improvement | Day 30, Month 3, Month 6, Month 9 and Month 12 after the first injection.
  Aesthetic improvement of the face will be assessed using the Global Aesthetic Improvement Scale, a 5-point scale ranking from 1: Very much improved to 5: worse. The lower the score, the better the aesthetic result. Assessed by subjects.
Investigator Global aesthetic improvement | Day 30, Month 3, Month 6, Month 9 and Month 12 after the first injection.
  Aesthetic improvement of the face will be assessed using the Global Aesthetic Improvement Scale, a 5-point scale a 5-point scale ranking from 1: Very much improved to 5: worse. The lower the score, the better the aesthetic result. Assessed by investigators.
Patient's quality of life | Day 30, Month 3, Month 6, Month 9 and Month 12 after the first injection.
  Quality of life will be assessed using Dermatology Life Quality Index (DLQI). The Dermatology Life Quality Index is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
  Assessed by subjects
Improvement of the patient's quality of life | Day 30, Month 3, Month 6, Month 9 and Month 12 after the first injection.
  Improvement will be assessed using a 4-point Likert scale (from 0-not improved to 3-Very much improved).
  Assessed by subject
Visual analogic scale pain assessment | Immediately after the injection (for initial injection only)
  Assessment of pain using a 0-100mm Visual Analogue Scale (0 corresponds to no pain and 100 corresponds to the highest pain that can be felt).
  Assessed by the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Maire, Principal Investigator — Centre Médical Saint-Jean
Locations (3):
- France (3):
  - Hôpital Roger Salengro, Lille, Nord
  - Cabinet médical, Toulouse, Occitanie
  - Cabinet médical, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No